CLINICAL TRIAL: NCT04792723
Title: Pharmacokinetic and Pharmacodynamic Study of a Novel Sublingual Aspirin Tablet Compared to Conventional Oral Aspirin in Healthy Subjects
Brief Title: Pharmacokinetic and Pharmacodynamic Study of a Novel Sublingual Aspirin Tablet
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vita Green Health Products Co. Ltd (Industry)
Responsible Party: Principal Investigator, Dr. Elaine Chow, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VG-BABE-19-01
Record Dates: First submitted 2021-03-04; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: single-dose, two-treatment, two-period, two-sequence, randomized, crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteer (Experimental): Sublingual or oral aspirin 80mg tablet, single dose, two-treatment, two-period, two-sequence, randomized, crossover design, with washout 1-2 weeks
  Interventions: Drug: Sublingual aspirin; Drug: Oral aspirin

INTERVENTIONS:
Drug: Sublingual aspirin — Vita Green Health Products sublingual aspirin 80 mg tablet
Drug: Oral aspirin — Synco (HK) oral aspirin 80mg tablet

SUMMARY:
The objective of the study is to compare the pharmacokinetics and pharmacodynamics of a new sublingual formulation of aspirin with that of oral aspirin when administered to healthy volunteers under fasting conditions. The test product is sublingual aspirin 80 mg manufactured by Vita Green Health Products Co. Ltd, Hong Kong and the reference product is oral aspirin 80mg tablet manufactured by Synco (HK) Ltd, Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

1. Male, 18 to 55 years of age
2. Body mass index between 18-27kg/m2
3. Accessible vein for blood sampling
4. High probability for compliance and completion of the study
5. No significant abnormalities in general physical examination
6. Subjects must agree to take effective contraceptive methods to prevent his partner pregnant during the time of first dose of study medication until one week of last dose administration

Exclusion Criteria:

1. History of hepatic, renal, biliary, cardiovascular, gastrointestinal, haematological and other chronic and acute diseases within 3 months prior to screening
2. Clinically relevant abnormality in physical examination, ECG evaluation, urine test, blood chemistry or haematological test at the discretion of the investigator
3. Positive results for hepatitis B at screening
4. Moderate smoker (on average more than 2 cigarettes a day within 1 month prior to the start of first dosing)
5. Moderate consumption of alcohol (on average more than one drink per day within 1 month prior to start of first dosing)
6. Blood donation of more than 350 ml within 4 weeks prior to start of first drug dosing
7. Treatment of aspirin within 4 weeks before first dosing
8. Volunteer in any other clinical drug study within 2 months prior to start of first dosing
9. Hypersensitivity to aspirin or other drug in its class

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-03-05 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Plasma-concentration time data of salicylic acid | pre dose and up to 24 hour post dose
  area under the plasma concentration-time curve from time zero to last measurable concentration time point for sublingual versus oral aspirin 80mg

SECONDARY OUTCOMES:
Peak plasma concentration of salicylic acid | pre dose and up to 24 hour post dose
  Peak plasma concentration for sublingual versus oral aspirin 80mg
Time to reach peak plasma concentration of salicylic acid | pre dose and up to 24 hour post dose
  Tmax of sublingual versus oral aspirin 80mg
Terminal phase elimination rate constant of salicylic acid | pre dose and up to 24 hour post dose
  Terminal phase elimination rate constant of sublingual versus oral aspirin 80mg
Terminal elimination half-life of salicylic acid | pre dose and up to 24 hour post dose
  Terminal elimination half-life of sublingual versus oral aspirin 80mg
Plasma concentration time data of thromboxane B2 | pre dose and up to 24 hour post dose
  Area under the curve for sublingual versus oral aspirin 80mg
Platelet aggregation by impedance aggregometry | pre dose and up to 360 minutes post dose
  Differences in platelet aggregation with sublingual versus oral aspirin 80mg

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Chow, Principal Investigator — Chinese University of Hong Kong